CLINICAL TRIAL: NCT04655677
Title: A Phase 1 Study Evaluating Safety and Efficacy of C-CAR039 Treatment in Subjects With Relapsed and/or Refractory NHL
Brief Title: A Study of C-CAR039 Treatment in Subjects With r/r NHL SubjectsNon-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Shanghai AbelZeta Ltd. (Industry)
Responsible Party: Principal Investigator, Yan Zhang, MD, Chief Physician, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0702-023
Record Dates: First submitted 2020-09-25; First posted 2020-12-07 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: B-cell Non-Hodgkin's Lymphoma
Keywords: CD19/CD20-directed CAR-T cells
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prizloncabtagene Autoleucel (Experimental): Prizlon-cel will be intravenously administered as a single infusion after lymphodepletion
  Interventions: Biological: Prizloncabtagene Autoleucel

INTERVENTIONS:
Biological: Prizloncabtagene Autoleucel — Autologous 2nd generation CD19/CD20-directed CAR-T cells, single infusion intravenously
  Other Names: C-CAR039

SUMMARY:
This is a single-center, open-label study to evaluate the safety and efficacy of C-CAR039 in relapsed and/or refractory B-NHL patients.

DETAILED DESCRIPTION:
The study will include the following sequential phases: Screening, Apheresis and C-CAR039 manufacturing, Baseline testing, Lymphodepleting, C-CAR039 infusion, and Follow-up Visit.

ELIGIBILITY:
Criteria: Inclusion Criteria:

1. Age 18-70 years (include 18 and 70), male or female;
2. Expected survival ≥ 12 weeks
3. ECOG score 0-2
4. CD19 or CD20 positive B-NHL confirmed by cytology or histology according to WHO2016 criteria, including DLBCL, PMBCL, tFL, FL and MCL
5. Relapsed or refractory disease after ≥ 2 lines (for FL, at least 3 lines) of standard therapy or relapsed after autologous stem cell transplantation (ASCT);
6. For CD20-positive subjects, they should have received at least one regimen containing anti-CD20-targeted therapy (such as rituximab). If they do not complete the regimen due to intolerance, the cause of intolerance should be recorded;
7. No contraindications of apheresis.
8. At least one measurable lesion according to Lugano 2014 criteria;
9. Adequate organ and bone marrow function
10. The patient volunteered to participate in the study and signed the Informed Consent.

Exclusion Criteria:

1. Malignant tumors other than diffuse large B-cell lymphoma, follicular lymphoma and mantle cell lymphoma within 5 years before screening, except fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical operation and breast ductal carcinoma in situ after radical operation;
2. Active HIV, HBV, HCV or treponema pallidum infection;
3. Any instability of systemic disease, including but not limited to active infection (except local infection), severe cardiac, liver, kidney, or metabolic disease need therapy
4. Any other uncontrolled active disease that hinders participation in the trial;
5. Any situation that the investigator believes would compromise the safety of the subject or interfere with the purpose of the study;
6. Female subjects who have been pregnant or breastfeeding, or who plan to conceive during or within 1 year after treatment, or male subjects' partner plans to conceive within 1 year after C-CAR039 infusion;
7. Active or uncontrolled infections requiring systemic treatment within 14 days before enrollment;
8. Patients who have previously been infected with tuberculosis.
9. Administered Corticosteroids and/or other immunosuppressants within 7 days before apheresis. and 5 days before the infusion of C-CAR039;
10. Patients with central nervous system involvement;
11. Any systemic antitumor therapy performed within 2 weeks before enrollment;
12. Those with medical conditions that prevent them from signing the written informed consent or from complying with the study procedures; or those who are unwilling or unable to comply with the study requirements;
13. Other conditions was considered unsuitable for enrollment by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Up to 24 months after C-CAR039 infusion
  Incidence and severity of adverse events after C-CAR039 infusion according to National Cancer Institute Common Terminology Criteria for Adverse Events v5.0 criteria

SECONDARY OUTCOMES:
Maximum concentration of C-CAR039 in the peripheral blood (Cmax) | Up to 24 Months after C-CAR039 infusion
  Detect CAR-T copies number by qPCR
Time to maximum concentration of C-CAR039 in the peripheral blood (Tmax) | Up to 24 Months after C-CAR039 infusion
  Detect CAR-T copies number by qPCR
Tlast of C-CAR039 in the peripheral blood after infusio (Tlast) | Up to 24 Months after C-CAR039 infusion
  Detect CAR-T copies number by qPCR
AUC0h-28d of C-CAR039 in the peripheral blood (AUC0-28d) | Up to 28 days after C-CAR039 infusion
  Detect CAR-T copies number by qPCR
Overall response rate (ORR) | Up to 24 Months after C-CAR039 infusion
  Complete response (CR) rate plus partial response (PR) rate by Lugano 2014 criteria
Duration of response (DOR) | Up to 24 Months after C-CAR039 infusion
  The time from the date of first response (PR or better) to the date of disease progression or death after C-CAR039 infusion
Progression-free survival (PFS) | Up to 24 Months after C-CAR039 infusion
  The time from C-CAR039 infusion to the date of progression as assessed by Lugano 2014 criteria or death
Overall survival (OS) | Up to 24 Months after C-CAR039 infusion
  The time from C-CAR039 infusion to the date of death

CONTACTS AND LOCATIONS:
Overall Officials: Daobin Zhou, PhD&MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing/China, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu W, Li P, Zhou L, Yang M, Ye S, Zhu D, Huang J, Yao X, Zhang Y, Li L, Zhao J, Zhu K, Li J, Zheng C, Lan L, Wan H, Yao Y, Zhang H, Zhou D, Jin J, Liang A. A phase 1 trial of prizloncabtagene autoleucel, a CD19/CD20 CAR T-cell therapy for relapsed/refractory B-cell non-Hodgkin lymphoma. Blood. 2025 Apr 3;145(14):1526-1535. doi: 10.1182/blood.2024026401. PMID 39813680